CLINICAL TRIAL: NCT01563445
Title: Multi-center, Phase II, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety and Preliminary Efficacy of Activated Recombinant Factor VII (NovoSeven®) for Preventing Early Hematoma Growth in Acute Intracerebral Hemorrhage (ICH)
Brief Title: Safety and Preliminary Efficacy of Activated Recombinant Human Factor VII for Preventing Early Hematoma Growth in Acute Intracerebral Haemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7ICH-2073
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Intracerebral Haemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- activated recombinant human factor VII (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — Subjects will be randomised to receive a single intravenous dose of either 5, 20, 40 and 80 mcg/kg body weight. Administered within the first 4 hours after the insult
  Arms: activated recombinant human factor VII
Drug: placebo — Subjects will be randomised to receive a single intravenous dose. Administered within the first 4 hours after the insult
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to evaluate the safety and preliminary efficacy of activated recombinant human factor VII (NovoSeven®) for preventing early hematoma growth in acute Intracerebral Hemorrhage (ICH).

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous ICH diagnosed by CT (Computerized Tomography) scanning within 3 hours of onset
* Signed informed consent form, or an exception from standard informed consent requirements

Exclusion Criteria:

* Time of onset of symptoms of ICH unknown or more than 3 hours prior to CT
* Patients with secondary ICH related to infarction, hemophilia or other coagulopathy, tumor, trauma, haemorrhagic infarction, cerebrovenous thrombosis, aneurysm, AVM (Arteriovenous Malformation) or severe trauma
* Surgical haematoma evacuation planned or performed within 24 hours of onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-11; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of a treatment-related serious adverse event (SAE)

SECONDARY OUTCOMES:
Occurrence of adverse events
Change in ICH volume as measured by CT head scans

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, New York, New York, United States

REFERENCES:
- [Result] Mayer SA, Brun NC, Broderick J, Diringer MN, Davis SM, Steiner T. Safety and Preliminary Efficacy of Recombinant Coagulation Factor VII in Patients with Acute Intracerebral Hemorrhage. Stroke 2004; 35: 322
- [Result] Diringer MN, Skolnick BE, Mayer SA, Steiner T, Davis SM, Brun NC, Broderick JP. Risk of thromboembolic events in controlled trials of rFVIIa in spontaneous intracerebral hemorrhage. Stroke. 2008 Mar;39(3):850-6. doi: 10.1161/STROKEAHA.107.493601. Epub 2008 Jan 31. PMID 18239180
- [Result] Mayer SA, Brun NC, Broderick J, Davis SM, Diringer MN, Skolnick BE, Steiner T; United States NovoSeven ICH Trial Investigators. Recombinant activated factor VII for acute intracerebral hemorrhage: US phase IIA trial. Neurocrit Care. 2006;4(3):206-14. doi: 10.1385/NCC:4:3:206. PMID 16757825
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com